CLINICAL TRIAL: NCT03574363
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy, Safety, and Pharmacokinetics of KBP-5074 in Patients With Moderate-to-Severe Chronic Kidney Disease and Uncontrolled Hypertension
Brief Title: Phase 2b Study of KBP-5074 in Subjects With Uncontrolled Hypertension and Advanced Chronic Kidney Disease
Acronym: BLOCKCKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBP5074-2-001
Record Dates: First submitted 2018-06-04; First posted 2018-07-02 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Hypertension
Keywords: Chronic Kidney Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — KBP-5074; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KBP-5074 0.25 mg tablet (Experimental): KBP-5074 0.25 mg tablet QD orally, 84 days
  Interventions: Drug: KBP-5074 0.25 mg tablet
- KBP-5074 0.5 mg tablet (Experimental): KBP-5074 0.5 mg tablet QD orally, 84 days
  Interventions: Drug: KBP-5074 0.5 mg tablet
- Placebo tablet (Placebo Comparator): Placebo tablet QD orally, 84 days
  Interventions: Drug: KBP-5074 0.25 mg tablet; Drug: KBP-5074 0.5 mg tablet

INTERVENTIONS:
Drug: KBP-5074 0.25 mg tablet — Oral administration, QD, 84 days
  Other Names: MRA
  Arms: KBP-5074 0.25 mg tablet; Placebo tablet
Drug: KBP-5074 0.5 mg tablet — Oral administration, QD, 84 days
  Other Names: MRA
  Arms: KBP-5074 0.5 mg tablet; Placebo tablet

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, multi-center study to assess the efficacy, safety, and pharmacokinetics of KBP-5074 in patients with moderate-to-severe chronic kidney disease and uncontrolled hypertension.

DETAILED DESCRIPTION:
The study will enroll up to 165 patients, randomized in a 1:1:1 ratio to 1 of 3 treatment groups (55 patients in each group): KBP-5074 0.25 mg once daily (QD), KBP-5074 0.5 mg QD, or placebo QD. Randomization will be stratified to balance enrollment for key variables that may influence safety and/or efficacy evaluations, including estimated Glomerular Filtration Rate (eGFR) (30 versus 29 mL/min/1.73 m2) and Systolic Blood Pressure (SBP) (160 versus <160 mmHg). The study will be approximately 5 months in duration with 84 days of double-blind treatment. The study will consist of an up to 4-week screening period; 2-week, open-label (placebo) run-in period; 84-day double-blind treatment period; and a 4-week post-treatment safety follow-up period. Patients will be sampled for plasma pharmacokinetics (PK). Total KBP-5074 levels will be assessed in patients treated with active drug. A total of 4 PK samples will be collected from each patient, including Day 1 (prior to discharge), Day 14 pre-dose, Day 28 pre-dose, and End of Study Visit (Day 98)/Early Termination Visit. The pre-dose samples assume that patients will be dosed in the unit on those days above. If patients are not dosed in the unit on those days, a flexible PK sample will be collected during each of these visits.Safety will be assessed systematically, and an independent data monitoring committee will perform cumulative reviews of safety data at regular intervals during the study. Serum potassium levels, serum creatinine, and blood pressure will be closely monitored throughout the study. At Screening, patients must have uncontrolled hypertension, defined as resting trough cuff seated SBP 140 mmHg, based on the mean of the last 2 consecutive blood pressure readings at Screening in the clinic. In all cases, dose and frequency of concurrent antihypertensive medications are expected to be maintained without change for 30 days prior to randomization in order to ensure that blood pressure is stable. In general, patients should not add nor adjust dose and/or types of the antihypertensive medications they are receiving during the screening period and throughout the duration of the study (unless they develop hypertensive crisis or symptomatic hypotension). Patients will be advised to maintain their normal diet and avoid alcohol or potassium-rich foods/drinks during the study period. No potassium supplements are permitted, unless clinically indicated to treat hypokalemia until serum potassium values are within the normal range. Potassium-sparing agents are not permitted. After completion of the screening period and the qualifying Screening Visit, patients who meet all eligibility criteria (except those criteria scheduled to be assessed after the Screening Visit), will enter the 2-week, open-label (placebo) run-in period. At the end of the run-in period, patients will be re-assessed for eligibility, including compliance to study drug received during the run-in period, which must be >80% and 120% (i.e. placebo and stable antihypertensive medication, i.e. no change in antihypertensive medication). If a patient is found to be ineligible during Screening, a 1-time re-screening is allowed if the Investigator believes that the patient's condition has changed and the patient may be eligible before the re-screening tests. Please note that a new patient number should be assigned to any re-screened patient, and all the procedures defined in the protocol for the Screening Visit and during the run-in period must be repeated. Patients who meet all eligibility criteria at the end of the screening period and run-in period will be randomized (stratified based on eGFR 30 versus 29 mL/min/1.73 m2 and SBP 160 versus <160 mmHg) into the study on Day 1. All randomized patients will receive double-blind treatment for 84 days. Patients will be followed for 4 weeks for safety assessments after the last dose of study drug. A subset of patients who still meet eligibility criteria at the end of the run-in period (Visit 3) will undergo 24-hour ambulatory blood pressure monitoring (ABPM) on Day 1, Day 40, and Day 82.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 85 years of age, inclusive. The lower age limit may be higher if it is legally required in the participating country;
2. Body mass index between 19 and 45 kg/m2, inclusive;
3. Stage 3B/4 CKD (defined as eGFR 15 and 44 mL/min/1.73 m2, based on the isotope dilution mass spectrometry traceable MDRD equation version 4, according to central laboratory results at Screening [single retest is allowed]);
4. Uncontrolled hypertension (Grade 1 to 2 systolic hypertension - ESC/ESH), defined as:

   * Resting trough cuff seated SBP 140 and 179 mmHg based on the mean of at least 2 current consecutive clinic blood pressure readings at Screening and at the end of the placebo run-in period (Visit 3); AND
   * Currently on 2 or more antihypertensive medications, which have been titrated upward as tolerated to recommended hypertension target doses (such as diuretics [except for potassium-sparing diuretics], renin angiotensin system blockers, and/or calcium channel blockers. One of the antihypertensive medications must be high ceiling diuretic (loop or thiazide like), unless there is a documented intolerance or contraindication to diuretic therapy. The doses of the antihypertensive medications should be stable without any dose adjustment during the 30 days prior to randomization; OR
   * Patients with uncontrolled hypertension and moderate-to-severe CKD with documented history of intolerance to multiple antihypertensive medications on fewer than 2 antihypertensive medications;
5. Serum potassium 4.8 mmol/L at both Screening and the end of the placebo run-in period. A single retest is allowed to exclude laboratory error or hemolyzed samples;
6. Women of childbearing potential (WOCBP) must agree to use 2 medically accepted, effective methods of birth control during the study and for 90 days after the end of the study. Adequate methods of contraception are defined as those that result in a low failure rate (< 1% per year) when used consistently and correctly. Such methods include the use of oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products (such as an intrauterine diaphragm, condoms, or spermicides);

   * WOCBP are defined as women who are not surgically or chemically sterilized, including hysterectomy or bilateral oophorectomy (tubal ligation is not acceptable), and who are between menarche and 1-year post-menopause; and
   * Post-menopausal is defined as amenorrheic for at least 1 year, AND if aged under 60 years, have a serum follicle-stimulating hormone (FSH) level > 20 mIU/L. Women who are taking hormone replacement therapy (HRT) do not have to have FSH assessments, but the amenorrhea (before starting HRT) must have been naturally (spontaneously) occurring and have been accompanied by an appropriate clinical profile (eg, age appropriate and history of vasomotor symptoms);
7. Males with partners who are WOCBP must agree to use condoms plus spermicide and their female partner must also be using contraception (eg, hormonal or intra-uterine device). This double contraception must be used from the first dose of study drug until at least 90 days after the last dose of study drug;
8. Males must also refrain from donating sperm during the study and for 90 days after the last dose; and
9. Capable of understanding the written informed consent, provide signed and witnessed written informed consent before any study-specific procedure, and agree to comply with protocol requirements.

Exclusion Criteria:

1. Resting trough seated SBP ≥180 or < 140 mmHg, based on the mean of at least 2 current consecutive clinic blood pressure readings at Screening and the end of the placebo run-in period (Visit 3);
2. Serum potassium > 4.8 mmol/L;
3. Compliance with medications (including both open-label placebo and current antihypertensive medications) < 80% or > 120% during the run-in period (assessed at Visit 3);
4. Currently on an MRA (eg, spironolactone or eplerenone) other than KBP-5074, or received any MRAs during the last 3 months prior to Screening, or currently on any potassium supplements;
5. Chronic or intermittent use of a potassium binder for the treatment of hyperkalemia from 3 months prior to Screening until the end of study assessments, including but not limited to calcium polystyrene sulfonates (eg, sorbisterit, calcium resonium), sodium polystyrene sulfonates (eg, kayexalate, anti-kalium sodium), and patiromer (eg, Veltassa™) and sodium zirconium cyclosilicate (eg, Lokelma™);
6. Have routinely or chronically used or required potassium-sparing diuretics (eg, amiloride, triamterene) within 3 months prior to Screening until the end of study assessments;
7. History of known/suspected contraindications, allergy, or intolerance to MRAs (eg, spironolactone, eplerenone) or has a known hypersensitivity to KBP-5074, other MRAs, or related compounds;
8. Clinically significant hyperkalemia while on an angiotensin converting enzyme inhibitor, angiotensin receptor blocker, direct renin inhibitor, and/or MRA, requiring down titration or discontinuation of above medication, or hospitalization for hyperkalemia within 3 months prior to Screening, or hyperkalemia > 5.6 mmol/L during the 2 weeks prior to Screening;
9. History/diagnosis of renal artery stenosis or history/diagnosis of renovascular hypertension;
10. Currently receiving HD, or peritoneal dialysis within 3 months prior to Screening, and those patients with an episode of acute kidney injury within 3 months of Screening;
11. History of a renal transplant, or impending renal transplant;
12. Acute decompensated heart failure including exacerbation of chronic heart failure manifested by signs and symptoms that may require hospitalization and/or intravenous diuretic therapy (New York Heart Association Class III to IV) within 3 months prior to Screening, or presence of hemodynamically significant valve diseases and/or other hemodynamically significant obstructive lesions of left ventricular outflow tract;
13. Major cardiac, cerebral, and/or carotid artery diseases, including but not limited to acute coronary syndrome, myocardial infarction, stroke, and/or transient ischemic attack; major cardiovascular or percutaneous procedures including cardiac ablation, coronary revascularization, and carotid angioplasty within 6 months prior to Screening; OR

    - Cardiovascular conditions likely to require surgical or percutaneous intervention within 6 months from Screening;
14. History of clinically significant arrhythmia, including but not limited to any of the following:

    * Symptomatic bradycardia and/or symptomatic ventricular arrhythmia within 3 months prior to Screening;
    * Second- or third-degree heart block; or
    * New onset or untreated atrial fibrillation; Note: Patients with stable (6 months) asymptomatic rate controlled atrial fibrillation on appropriate therapy, which may include anticoagulation, are permitted.
15. QT interval corrected using Fridericia's formula (QTcF) > 450 ms for males or > 470 ms for females at Screening or Day 1; QTcF should be the average of the required triplicate set of ECGs at each timepoint;
16. History of prolonged QT interval;
17. History or family history of sudden cardiac death or long QT syndrome;
18. History of cardiac transplant, on a heart transplant list, or has a left ventricular assistance device;
19. History of clinically significant acute or chronic hepatitis (including infectious, metabolic, autoimmune, genetic, ischemic, or other forms), hepatocirrhosis, or hepatic tumors;
20. History of gastrointestinal surgery that might affect absorption/oral bioavailability of oral antihypertensive therapies including KBP-5074;
21. Clinically significant abnormal liver function test at Screening or the end of the run-in period (Visit 3), defined as aspartate aminotransferase or alanine aminotransferase > 3 × the upper limit of normal (ULN) or total bilirubin > 2 × ULN;

    * Note: Patients with total bilirubin > 2 × ULN and history of Gilbert's syndrome may be included.
22. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) antibody;
23. History of malignancy in the past 5 years, with the exception of basal or resected cutaneous squamous cell carcinoma of the skin or carcinoma in situ, prostate cancer in situ with a normal prostate-specific antigen post treatment, cervical carcinoma in situ, gastric cancer in situ, colon cancer in situ adequately treated with no progression over the past 2 years;
24. History of prescription drug abuse, illicit drug use, or alcohol abuse according to medical history within 6 months prior to Screening;
25. A positive drug screen test (excluding a positive result secondary to a prescribed medication from a physician, or tetrahydrocannabinol) at Screening or the end of the run-in period (Visit 3);
26. Female patients who are known to be pregnant or breastfeeding;
27. Previously enrolled in any KBP-5074 study;
28. Receipt of any other investigational product within 30 days or 5 half-lives (whichever is longer) prior to Screening;
29. Use of any nutrients known to modulate cytochrome P450 (CYP)3A activity (based on the KBP-5074 metabolic pathway) or any strong or moderate inhibitors or inducers of CYP3A4, starting from 14 days prior to the first dose of study drug at Day 1 until the end of study assessments, including but not limited to the following: inhibitors, such as ketoconazole, miconazole, itraconazole, fluconazole, atazanavir, erythromycin, clarithromycin, ranitidine, and cimetidine, and inducers, such as rifampicin, rifabutin, glucocorticoids, carbamazepine, phenytoin, phenobarbital, and St. John's wort;
30. Has donated or lost a significant volume (> 500 mL) of blood or plasma within 30 days prior to Screening;
31. An employee or family member of the Investigator or study site personnel;
32. Unlikely to comply with the protocol requirements, instructions, and/or study-related restrictions (eg, uncooperative attitude, unavailable for follow up call, and/or improbability of completing the clinical study); and
33. History of any other prior or concomitant clinical condition or acute and/or unstable systemic disease not listed above that, in the opinion of the Investigator, compromises patient inclusion, such as a history or presence of clinically decompensated or unstable cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, or concomitant morbidity of such severity that the patient is likely to die within 1 year from Screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - KBP Biosciences USA Inc, Princeton, New Jersey
  - Worldwide Clinical Trials, Morrisville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakris G, Pergola PE, Delgado B, Genov D, Doliashvili T, Vo N, Yang YF, McCabe J, Benn V, Pitt B; BLOCK-CKD Study Group. Effect of KBP-5074 on Blood Pressure in Advanced Chronic Kidney Disease: Results of the BLOCK-CKD Study. Hypertension. 2021 Jul;78(1):74-81. doi: 10.1161/HYPERTENSIONAHA.121.17073. Epub 2021 May 10. PMID 33966452
- [Derived] Bakris G, Yang YF, Pitt B. Mineralocorticoid Receptor Antagonists for Hypertension Management in Advanced Chronic Kidney Disease: BLOCK-CKD Trial. Hypertension. 2020 Jul;76(1):144-149. doi: 10.1161/HYPERTENSIONAHA.120.15199. Epub 2020 Jun 10. PMID 32520623

RESULTS

PARTICIPANT FLOW:
Groups:
- KBP-5074 .25mg: KBP-5074 low dose
- KBP-5074 .5mg: KBP-5074 high dose
- Placebo: Placebo to match active drug
Period: Overall Study
Arm/Group | KBP-5074 .25mg | KBP-5074 .5mg | Placebo
Started | 51 | 54 | 57
Completed | 47 | 44 | 47
Not Completed | 4 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KBP-5074 .25mg | KBP-5074 .5mg | Placebo | Total
Number analyzed (Participants) | 51 | 54 | 57 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 27 | 74
  >=65 years | 28 | 30 | 30 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 23 | 73
  Male | 24 | 31 | 34 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 15 | 35
  Not Hispanic or Latino | 39 | 46 | 42 | 127
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 2 | 12
  White | 46 | 49 | 54 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  North America | 18 | 18 | 20 | 56
  Europe | 31 | 34 | 36 | 101
  Chile | 1 | 2 | 0 | 3
  Israel | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Change in trough cuff resting seated SBP from baseline to Day 84.
Time Frame: Baseline to Day 84
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo Tablet | KBP-5074 0.25 mg Tablet | KBP-5074 0.5 mg Tablet
Number analyzed (Participants) | 57 | 51 | 54
mmHg
  Baseline | 155.8 (1.44) | 154.3 (2.11) | 155.7 (2.01)
  Day 84 | 150.4 (1.98) | 142.8 (2.65) | 139.9 (2.65)
  Change from Baseline to Day 84 | -5.3 (2.39) | -11.5 (2.9) | -15.9 (3.15)

2. Secondary Outcome: Diastolic Blood Pressure
Description: Change in trough cuff seated DBP from baseline to Day 84
Time Frame: Baseline to Day 84
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo Tablet | KBP-5074 0.25 mg Tablet | KBP-5074 0.5 mg Tablet
Number analyzed (Participants) | 57 | 51 | 54
mmHg
  Baseline | 85.9 (1.52) | 89 (1.7) | 88.4 (1.78)
  Day 84 | 83.8 (1.34) | 82.2 (1.68) | 81.4 (1.90)
  Change from Baseline to Day 84 | -2.0 (1.41) | -6.7 (2.02) | -7.0 (2.23)

3. Secondary Outcome: UACR
Description: Change in UACR from baseline to Day 84
Time Frame: Baseline to Day 84
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Placebo Tablet | KBP-5074 0.25 mg Tablet | KBP-5074 0.5 mg Tablet
Number analyzed (Participants) | 43 | 36 | 44
mg/g
  Baseline | 483.7038 [288.6661 to 810.5189] | 700.4447 [465.8093 to 1053.2694] | 519.0621 [328.9336 to 819.0876]
  Day 84 | 313.91930 [160.8878 to 612.5096] | 435.7897 [256.8354 to 739.4333] | 372.0062 [217.4223 to 636.4968]
  Change from Baseline to Day 84 | 0.6927 [0.4868 to 0.9858] | 0.6222 [0.3590 to 1.0781] | 0.7328 [0.4774 to 1.1249]

4. Other Pre Specified Outcome: Total KBP-5074 Concentration
Description: Total KBP-5074 concentration
Time Frame: Day 84
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE collection started with the signing of the ICF followed by 4 weeks of screening period, then 2 weeks of run-in period, then 84 days of double-blind study treatment, then 4 weeks of safety follow up. Total AE collection period was 22 weeks.
Arm/Group | Placebo Tablet | KBP-5074 0.25 mg Tablet | KBP-5074 0.5 mg Tablet
All-Cause Mortality (participants affected / at risk) | 2/57 | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 4/57 | 1/51 | 2/54
Other Adverse Events (participants affected / at risk) | 15/57 | 20/51 | 34/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablet (N=57) | KBP-5074 0.25 mg Tablet (N=51) | KBP-5074 0.5 mg Tablet (N=54)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) — unknown cause
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablet (N=57) | KBP-5074 0.25 mg Tablet (N=51) | KBP-5074 0.5 mg Tablet (N=54)
Hyperkalemia (Metabolism and nutrition disorders) | 14 (26) | 15 (33) | 28 (52)
CKD (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
eGFR decrease (Investigations) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results are only unblinded after full study is completed. Therefore, PI would be unable to disclose results until after the full database lock and unblinding.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03574363/Prot_SAP_000.pdf